CLINICAL TRIAL: NCT01292590
Title: Use of Closed Loop Control to Examine the Effect of Changes in Dietary Fat Intake on Insulin Requirements and Glucose Control
Brief Title: Effect of Dietary Fat on Glycemic Control in Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Joslin Diabetes Center (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-P-000140/1; BIDMC
Record Dates: First submitted 2010-10-21; First posted 2011-02-09 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Nutrients

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- High fat meal (Experimental)
  Interventions: Other: High fat meal

INTERVENTIONS:
Other: High fat meal — 40 grams saturated fat
  Other Names: Macronutrient

SUMMARY:
The purpose of this study is to determine if dietary fat alters insulin requirements in type 1 diabetes.

DETAILED DESCRIPTION:
This cross-over prospective study will require a two day admission to the clinical research center. Subjects will undergo closed loop glucose control and will received a diet with controlled macronutrient content.

ELIGIBILITY:
Inclusion Criteria:

* type 1 diabetes using insulin pump and CGM

Exclusion Criteria:

* renal or hepatic failure
* cancer or lymphoma
* malabsorption or malnourishment
* hypercortisolism
* alcoholism or drug abuse
* anemia (hematocrit < 36 in females and <40 in males)
* eating disorder
* dietary restrictions
* Acetaminophen allergy
* Chronic acetaminophen use
* Glucocorticoid therapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-09; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Change in insulin requirements | postprandially until 8 hours

CONTACTS AND LOCATIONS:
Overall Officials: Howard Wolpert, MD, Principal Investigator — Joslin Diabetes Center/Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States